CLINICAL TRIAL: NCT01822756
Title: A Phase 1b Study of the Safety and Tolerability of Ruxolitinib in Combination With Gemcitabine With or Without Nab-Paclitaxel in Subjects With Advanced Solid Tumors
Brief Title: An Open-Label Study of Ruxolitinib Given With Chemotherapy in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Dose escalation ended after Cohort B1, RUX 10 mg BID - GCSF in October 2014.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-144
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — ruxolitinib; Gemcitabine; 130-nm albumin-bound paclitaxel; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A -ruxolitinib, gemcitabine (Experimental): Ruxolitinib (RUX) was self-administered by the subject orally in the morning and evening, approximately 12 hours apart, without regard to food. The morning dose of RUX was to be taken before the chemotherapy infusion, Gemcitabine IV, on days when they were given together (Days 1, 8, and 15 of each cycle).
  Interventions: Drug: ruxolitinib; Drug: gemcitabine
- Regimen B-ruxolitinib, gemcitabine, nab-paclitaxel, filgrastim (Experimental): Ruxolitinib (RUX) was self-administered by the subject orally in the morning and evening, approximately 12 hours apart, without regard to food.
  Gemcitabine was provided as open-label, commercial product and was administered intravenously (IV) over 30 minutes on Days 1, 8, and 15 of each 28-day cycle. Reduced doses of gemcitabine administered IV over 30 minutes on Days 1, 8, and 15 of each 28-day cycle could also be explored.
  nab-Paclitaxel, as open-label, commercial product, was administered IV over 30 minutes on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: ruxolitinib; Drug: gemcitabine; Drug: nab-paclitaxel; Drug: filgrastim

INTERVENTIONS:
Drug: ruxolitinib
Drug: gemcitabine — Other names: Gemzar®
Drug: nab-paclitaxel — Other names: Abraxane®
  Arms: Regimen B-ruxolitinib, gemcitabine, nab-paclitaxel, filgrastim
Drug: filgrastim — Prophylactic GCSF support was filgrastim and was given in Cycle 1 on Days 2 to 5, 9 to 12, and 16 to 19, unless chemotherapy was held for toxicity, then prophylactic GCSF support was also held.
  Other Names: Neupogen®
  Arms: Regimen B-ruxolitinib, gemcitabine, nab-paclitaxel, filgrastim

SUMMARY:
This is a study of ruxolitinib in combination with gemcitabine with or without nab-paclitaxel administered to patients with advanced or metastatic pancreatic cancer. The study will be conducted in two parts.

Part 1 of the study will evaluate the safety, tolerability and pharmacokinetics (PK) of ruxolitinib when given as described to patients with advanced or metastatic pancreatic cancer. A goal of Part 1 will be to identify the maximally tolerated dose (MTD) of ruxolitinib when given with gemcitabine with or without nab-paclitaxel. This dose will be selected for use in Part 2 of the study.

Part 2 of the study will further evaluate the safety, tolerability, PK and preliminary clinical activity of ruxolitinib at the dose defined in Part 1 used in combination with gemcitabine with or without nab-paclitaxel in subjects with advanced or metastatic pancreatic cancer.

After multiple challenges of trial conduct, by mutual agreement between investigators and sponsor, dose escalation ended after Cohort B1, RUX 10 mg twice daily (BID) - GCSF in October 2014. Therefore, the MTD was not reached. No safety issues led to the decision to stop further enrollment.

Because of the early study termination, samples for pharmacokinetics and pharmacodynamics, and computed tomography for tumor burden were collected, but not analyzed; analysis data are not available. The data cutoff for this posting is 22 SEP 2015. As of the data cutoff, 1 subject was receiving treatment in the study and had been enrolled for 47 weeks. This subject had their end of treatment visit in AUG 2016. A comparison of this subjects' safety data after the cutoff date showed no clinically meaningful differences (eg, adverse events) compared with safety results that are summarized here.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older
* Histologically or cytologically confirmed adenocarcinoma of the pancreas
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Requirements for prior therapy as outlined below:

  * Enrollment into Regimen A: received no more than 1 prior chemotherapy regimen for advanced or metastatic disease (not including neoadjuvant and/or adjuvant therapy)
  * Enrollment into Regimen B: received no prior chemotherapy for advanced or metastatic disease (not including neoadjuvant and/or adjuvant therapy)
* Adequate renal, hepatic, and bone marrow function without blood product or hematopoietic growth factor support:
* Able to swallow and retain oral medication

Exclusion Criteria:

* Any known contraindications to the use of gemcitabine (for enrollment in Regimen A or B) or nab-paclitaxel (for enrollment into Regimen B).
* Evidence of uncontrolled brain metastases or history of uncontrolled seizures.
* Ongoing radiation therapy and/or radiation therapy administered within 28 days of enrollment. Subjects who have received radiation to the spine, pelvis, ribs, or femur should be discussed with the sponsor, as extensive radiation to marrow forming region may compromise a subject's ability to tolerate myelosuppressive chemotherapy. Subjects who have ongoing radiotherapy-related toxicities are not eligible.
* Subjects who participated in any other study in which receipt of an investigational study drug occurred within 28 days or 5 half-lives (whichever is longer) prior to first dose.
* Current or previous other malignancy within 2 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or other noninvasive malignancy without sponsor approval.
* Inability to swallow food or any condition of the upper GI tract that precludes administration of oral medications.
* Recent (≤ 3 months) history of partial or complete bowel obstruction.
* Unwilling to be transfused with blood components.
* Known history of Hepatitis B or C infection or HIV infection.
* Presence of ≥ Grade 2 neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2015-09 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fitzroy Dawkins, M.D., Study Director — Incyte Corporation
Locations (5):
- United States (5):
  - Birmingham, Alabama
  - Gainesville, Florida
  - Sarasota, Florida
  - Durham, North Carolina
  - Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A0: RUX 15 mg BID; Gemcitabine 1000 mg/m^2 on Days 1, 8, and 15
- Cohort B (-1): RUX Orally, Twice Daily 5 mg BID; Gemcitabine 1000 mg/m^2 on Days 1, 8, and 15; nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15; + GCSF
- Cohort B0 (+GCSF): RUX 10 mg BID; Gemcitabine 1000 mg/m^2; nab-Paclitaxel 100 mg/m^2; +GCSF
- Cohort B0 (-GCSF): RUX 10 mg BID; Gemcitabine 1000 mg/m^2; nab-Paclitaxel 100 mg/m^2; -GCSF
- Cohort B1: RUX 10 mg BID; Gemcitabine 1000 mg/m^2; nab-Paclitaxel 100 mg/m^2; - GCSF given in Cycle 1 on Days 2 to 5, 9 to 12, and 16 to 19
Period: Overall Study
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Started | 16 | 4 | 10 | 4 | 8
Discontinued From the Study | 16 | 4 | 10 | 4 | 7
Completed | 0 | 0 | 0 | 0 | 1
Not Completed | 16 | 4 | 10 | 4 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0
Not completed — Disease progression | 11 | 1 | 7 | 2 | 6
Not completed — Death | 2 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0
Not completed — disease progression & patient preference | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Subjects (ITT): All subjects who received at least 1 dose of Ruxolitinib (RUX).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1 | Total
Number analyzed (Participants) | 16 | 4 | 10 | 4 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (8.56) | 61.3 (6.40) | 61.2 (9.33) | 70.0 (7.62) | 62.4 (8.48) | 62.8 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 6 | 0 | 2 | 20
  Male | 8 | 0 | 4 | 4 | 6 | 22
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Graded from 0- 2; 0 being fully active, able to carry on all pre-disease performance without restriction 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature and 2 Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours.
  participants
    0 | 6 | 2 | 8 | 3 | 5 | 24
    1 | 10 | 2 | 2 | 1 | 3 | 18
    2 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events That Are Defined as Dose Limiting Toxicities (DLTs)
Description: Toxicities occurring during the first treatment cycle (Cycle 1) defined tolerability. Within each cohort, subjects were considered evaluable if they had received at least 40 of 56 planned doses of RUX during the 28-day surveillance period and received 2 of the 3 planned doses of chemotherapy (gemcitabine and/or gemcitabine and nab-paclitaxel) at the assigned dose level, or they had experienced a DLT.
Time Frame: Approximately 28 days
Population: Safety population included all enrolled subjects who received at least 1 dose of RUX.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 16 | 4 | 10 | 4 | 8
percentage of participants | 0.0 | 0.0 | 20.0 | 50.0 | 0.0

2. Secondary Outcome: Plasma Concentrations Will be Used to Estimate Peak Plasma Concentration (Cmax) and Area Under the Plasma Concentration Curve (AUC).
Time Frame: Day 1 and Day 8
Population: Further enrollment of additional study cohorts was stopped after Cohort B1, RUX 10 mg BID - GCSF; Part 2 of the study was not conducted. Because of the early study termination, samples for pharmacokinetics and pharmacodynamics, and computed tomography for tumor burden were collected, but not analyzed; analysis data are not available.
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Plasma Concentration of Tumor Specific Biomarkers and Cytokines Before and During Treatment.
Time Frame: Up to 6 months
Population: Enrollment of additional study cohorts was stopped after Cohort B1, RUX 10 mg BID-GCSF; Part 2 of the study was not conducted.Because of the early study termination, samples for pharmacokinetics and pharmacodynamics, and computed tomography for tumor burden were collected, but not analyzed; analysis data are not available.
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Clinical Activity as Measured by the Greatest Decrease in Tumor Burden Compared to Baseline.
Time Frame: Approximately 6 months
Population: Enrollment of additional study cohorts was stopped after Cohort B1, RUX 10 mg BID-GCSF; Part 2 of the study was not conducted. Because of the early study termination, samples for pharmacokinetics and pharmacodynamics, and computed tomography for tumor burden were collected, but not analyzed; analysis data are not available.
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With a Best Response by RECIST Criteria
Description: Best response was determined on the subject level using the highest overall response achieved post-baseline. In the case of stable disease (SD), measurements had to meet the SD criterion at least once after study entry at a minimum interval of 49 days. Subjects who failed to meet this criterion had best response of progressive disease (PD) if the next available RECIST evaluation after the initial scan indicated PD or not evaluable (NE) if no additional RECIST evaluations were available.
  Complete Response (CR) and Partial Response (PR) defined by the Response Evaluation Criteria in Solid Tumor (RECIST) criteria. CR: Disappearance of all target and nontarget lesions. PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter, or persistence of 1 or more nontarget lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: every 2 cycles starting at Cycle 3 Day 1 up to approximately 4 to 6 months
Population: Intent-to-Treat (ITT) Population - All subjects who received at least 1 dose of RUX
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 16 | 4 | 10 | 4 | 8
percentage of participants
  Overall response | 12.5 | 25.0 | 50.0 | 25.0 | 37.5
  Complete response | 0.0 | 0.0 | 0.0 | 25.0 | 0.0
  Partial response | 12.5 | 25.0 | 50.0 | 0.0 | 37.5
  Stable disease | 25.0 | 75.0 | 20.0 | 50.0 | 25.0
  Progressive disease | 37.5 | 0.0 | 10.0 | 0.0 | 37.5
  Not evaluable | 6.3 | 0.0 | 0.0 | 0.0 | 0.0
  Missing | 18.8 | 0.0 | 20.0 | 25.0 | 0.0

6. Secondary Outcome: Percentage of Responders
Description: Duration of response was measured as the time from the first overall response contributing to an objective response to the first overall response of progressive disease (PD) occurring after the first overall response contributing to the objective response.
Time Frame: Randomization to clinical cutoff 22Sept2015 (approx 244 days)
Population: Intent-to-Treat Population (ITT) population - All subjects who received at least 1 dose of RUX
Measure: Number; unit: Percentage of responders
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 16 | 4 | 10 | 4 | 8
Percentage of responders | 12.5 | 25.0 | 50.0 | 25.0 | 37.5

7. Secondary Outcome: Duration of Response
Description: Duration of response was the time from the first overall response contributing to an objective response to the first overall response of progressive disease (PD) occurring after the first overall response contributing to the objective response. Confidence intervals for median duration of response were calculated using the method of Brookmeyer and Crowley (1982).
Time Frame: Randomization to clinical cutoff 22Sept2015 (approx 244 days)
Population: Intent-to-Treat Population (ITT) population - All subjects who received at least 1 dose of RUX
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Number analyzed (Participants) | 16 | 4 | 10 | 4 | 8
days | 132.0 [NA to NA] — Not estimated; insufficient number of participants with events. | 33.0 [NA to NA] — Not estimated; insufficient number of participants with events. | 113.0 [57.0 to 533.0] | 244.0 [NA to NA] — Not estimated; insufficient number of participants with events. | 225.0 [57.0 to 225.0]

ADVERSE EVENTS:
Time Frame: From randomization to 30 days after last visit up to approximately 6 months.
Description: Safety population included all enrolled subjects who received at least 1 dose of RUX.
Arm/Group | Cohort A0 | Cohort B (-1) | Cohort B0 (+GCSF) | Cohort B0 (-GCSF) | Cohort B1
Serious Adverse Events (participants affected / at risk) | 10/16 | 4/4 | 3/10 | 0/4 | 2/8
Other Adverse Events (participants affected / at risk) | 16/16 | 4/4 | 10/10 | 4/4 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A0 (N=16) | Cohort B (-1) (N=4) | Cohort B0 (+GCSF) (N=10) | Cohort B0 (-GCSF) (N=4) | Cohort B1 (N=8)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hyperbilirubinemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Eye infection toxoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngeal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A0 (N=16) | Cohort B (-1) (N=4) | Cohort B0 (+GCSF) (N=10) | Cohort B0 (-GCSF) (N=4) | Cohort B1 (N=8)
Anaemia (Blood and lymphatic system disorders) | 9 | 2 | 6 | 4 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 2 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 1 | 6 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 5 | 1 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 8 | 2 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2 | 5 | 0 | 0
Chills (General disorders) | 1 | 0 | 1 | 1 | 1
Fatigue (General disorders) | 10 | 4 | 8 | 2 | 5
Feeling jittery (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 4 | 3 | 5 | 2 | 4
Pyrexia (General disorders) | 5 | 1 | 4 | 1 | 1
Haemobilia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 3 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0 | 5
Platelet count decreased (Investigations) | 3 | 0 | 1 | 0 | 2
White blood cell count decreased (Investigations) | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 2 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 2 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 1 | 2 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 4 | 2 | 4
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 3 | 0 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1 | 2
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 3 | 0 | 0
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0
Catheter site rash (General disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0
Local swelling (General disorders) | 0 | 1 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Cardiac enzymes increased (Investigations) | 0 | 0 | 1 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 3 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 2 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 2
White blood cell count increased (Investigations) | 0 | 0 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1 | 2 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 3 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 7 | 1 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Colonic Polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
In October 2014, further enrollment of additional study cohorts was stopped; Part 2 of the study wasn't conducted. Pharmacokinetic and Pharmacodynamics analyses weren't performed due to early termination. Maximum tolerated dose (MTD) was not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.